CLINICAL TRIAL: NCT01980446
Title: Cognitive Auditory Evoked Potential After Cardiac Arrest: Interest of Mismatch negativiTY: The CAPACITY Study
Brief Title: Cognitive Auditory Evoked Potential After Cardiac Arrest: Interest of Mismatch negativiTY
Acronym: CAPACITY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: P091118; 2010-A01378-31 (Other: IDRCB)
Record Dates: First submitted 2013-10-24; First posted 2013-11-11 (Estimated); Last update posted 2020-08-20 (Actual); Status verified 2020-08

CONDITIONS: Coma; Cardiac Arrest
Keywords: Coma; Cardiac arrest; Neurophysiology; Auditory evoked potential
MeSH Terms: conditions — Coma; Heart Arrest | interventions — Evoked Potentials, Auditory

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1:Mismatch negativity (Other): Presence of the mismatch negativity during the cortical auditory-evoked potential would predict a favorable outcome in comatose survivors after cardiac arrest.
  Interventions: Procedure: Auditory-evoked potentials

INTERVENTIONS:
Procedure: Auditory-evoked potentials — cortical auditory-evoked potentials are performed to all included patients at inclusion, at day 5 to day 10, day without sedation (up to 1 year), day of awakening

SUMMARY:
Determination of vital and functional outcome in comatose survivors after cardiac arrest is principally based on the identification of predictors of non-awakening, using by clinical, biological and electrophysiological tools. In patients without presence of non-awakening predictors, it would be of interest to identify predictive criteria of awakening. The presence of mismatch negativity during the cortical auditory-evoked potential could contribute to further progress in neurological prognostication of these patients. However, at this time, its prognostic value has been insufficiently studied and the optimal time of realization remains unknown.

DETAILED DESCRIPTION:
We hypothesized that the presence of the mismatch negativity during the cortical auditory-evoked potential would predict a favorable outcome in comatose survivors after cardiac arrest.The main objective is to determine the capacity of the presence of the mismatch negativity during the cortical auditory-evoked potential to predict a 1-year favorable outcome in comatose survivors after cardiac arrest

The secondary objectives are:

* To assess the capacity of the presence of the mismatch negativity during the cortical auditory-evoked potential to predict awakening during the hospitalisation stay.
* To determine the optimal time of realization of the cortical auditory-evoked potential
* To determine the capacity of the presence of the mismatch negativity during the cortical auditory-evoked potential to predict ICU discharge and/or hospital discharge favorable outcome in comatose survivors after cardiac arrest
* To determine the impact of the sedations drugs during the hypothermia phase, and during the ICU stay The main judgement criterion is the 1-year CPC score (CPC 1 to 2 as a favorable outcome)

Study design : Prospective, multicentre, interventional study. Decision making to withdrawal of life support will be strictly codified according current knowledge and standardized among the participating centres. In the absence of predictors of non-awakening, care will be continued without limitation. The design of the study will focus on the determination of the capacity of the presence of the mismatch negativity during the cortical auditory-evoked potential to predict awakening. Cortical auditory-evoked potential will be performed bedside in the ICU by qualified neurophysiologists. Results of cortical auditory-evoked potential will remain blinded of bedside clinicians providing care for the patients. Awakening will be assessed bedside daily. CPC score will be evaluated at discharge of the ICU, of the hospital, at 3 months and 1 year by an independent evaluator, blinded of the results of the cortical auditory-evoked potentials.

ELIGIBILITY:
Inclusion Criteria:

* Adults (age ≥ 18 years)
* hospitalized in the intensive care unit in the aftermath of a intra-or extra-hospital cardiac arrest
* alive but remaining comatose between the 2nd day and the 5th day after cardiopulmonary arrest

Exclusion Criteria:

* moribund patients (treatment limitations or the life expectancy of the inclusion estimated at less than 1 year)
* patient awake at day of potential inclusion
* brain death state
* failure to realize the cortical
* patient whose hearing loss is known

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
CPC score of 1 or 2 (favorable outcome) | 1 year
  1-year CPC score of 1 or 2 (favorable outcome)

SECONDARY OUTCOMES:
Awakeness | up to 1 year
  Awakeness during the hospitalisation stay
Time of realization of the cortical auditory-evoked potential | up to 1 year
  the optimal time of realization of the cortical auditory-evoked potential
CPC score of 1 or 2 at ICU discharge | up to 1 year
  the CPC score of 1 or 2 at ICU and at hospital discharge
Length of mechanical ventilation, ICU stay, hospital stay and vital status at discharge | up to 1 year
  impact of the sedations drugs during the ICU stay impact of therapeutic hypothermia
CPC score of 1 or 2 at hospital discharge | up to 1 year
  the CPC score of 1 or 2 at hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Stephane LEGRIEL, MD, Principal Investigator — Versailles Hospital - 78150 Le Chesnay - France
Locations (2):
- France (2):
  - Lariboisière Hospital - Medical and toxicology unit, Paris
  - Dr Stéphane LEGRIEL - Intensive Care Unit, Versailles